CLINICAL TRIAL: NCT05367934
Title: The Effect of Therapeutic Treatment Applied to Nursing Students on Perceived Stress and Stress Coping Behaviors: A Randomized Controlled Experimental Study
Brief Title: The Effect of Therapeutic Treatment on Stress and Coping Stress
Acronym: nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zehra Bayram (Other)
Responsible Party: Sponsor-Investigator, Zehra Bayram, Nurse, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0001-9237-2714
Record Dates: First submitted 2022-04-27; First posted 2022-05-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Nurse's Role
Keywords: nursing, therapeutic touch, stress, coping stress, education
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental study.
Who Masked: Participant
Masking Description: The nurses in the intervention group were given therapeutic touch for 15 minutes once a week for two weeks, and the patients in the control group did not receive any treatment other than their routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Therapeutic Touch on Nursing Students on Perceived Stress and Stress Coping Behaviors (Experimental): The nurses in the intervention group were given therapeutic touch for 15 minutes once a week for two weeks.
  Interventions: Behavioral: Therapeutic Touch
- The Effect of Therapeutic Touch on Stress and Stress Coping Behaviors (Other): No treatment was applied to the patients in the control group other than their routine care.
  Interventions: Behavioral: Therapeutic Touch

INTERVENTIONS:
Behavioral: Therapeutic Touch — Therapeutic Touch for stress

SUMMARY:
Nursing students are exposed to intensive theoretical and clinical applications throughout their academic education. During this educational process, students' stress increases and their coping behaviors are affected.

DETAILED DESCRIPTION:
This study was conducted to determine the effects of therapeutic touch applied to nursing students on stress levels and coping behaviors. The nurses in the intervention group were given therapeutic touch for 15 minutes once a week for two weeks, and the patients in the control group did not receive any treatment other than their routine care.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18, Maximum age 24 Volunteer to work, Nursing students who had not received touch therapy before were included in the study.

Exclusion Criteria:

* • Previous or current tactile therapy,

  * A therapeutic touch therapist,
  * Nursing students who did not volunteer for the study were not included in the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
The Effect of Therapeutic Touch on Stress | Scales are filled after 3 days of application
  Perceived Stress Inventory for Nursing Students (APPS) (Annex II) Sheu et al. (2002) originally in Chinese, the scale consisted of 29 items. Chan et al. (2009), Cronbach's alpha coefficient was found to be 0.89, and the sub-dimensions were 0.87-0.89. Karaca et al. (2014) validated the Turkish validity and reliability of the scale. In the evaluation of the items; A five-point Likert-type assessment was used, including '4- Very stressful for me, 3, 2, 1, 0- Not stressful for me'.
The Effect of Therapeutic Touch on Stress Coping Behaviors | Scales are filled after 3 days of application
  Stress Coping Behaviors Scale for Nursing Students (SPSAS) (Annex III), Sheu et al. (2002) the scale consists of 19 items. Karaca et al. (2014) validated the Turkish validity and reliability of the scale. Cronbach's alpha coefficient was found to be 0.76. In the evaluation of the items; A five-point Likert-type assessment was used: '4- I agree, 3, 2, 1, 0- I strongly disagree'.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Kuşçu Karatepe, phD, Principal Investigator — Osmaniye Korkut Ata University
Locations (1):
- Zehra Bayram, Osmaniye, Turkey (Türkiye)